CLINICAL TRIAL: NCT03753074
Title: A Multinational, Multicenter, Open-label, Randomized Controlled Trial to Investigate the Effectiveness of Tenofovir Alafenamide in Reducing Clinical Events in Chronic Hepatitis B Patients Beyond Treatment Indications by Current Guidelines
Brief Title: Effectiveness of TAF in Reducing Clinical Events in CHB Patients Beyond Treatment Indications by Current Guidelines
Acronym: ATTENTION
Status: Active, not recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Young-Suk Lim (Other)
Collaborators: Samsung Medical Center (Other); Kyunghee University Medical Center (Other); Chung-Ang University Hosptial, Chung-Ang University College of Medicine (Other); Seoul National University Hospital (Other); Ulsan University Hospital (Other); Konkuk University Medical Center (Other); Kyungpook National University Hospital (Other); Korea University Guro Hospital (Other); Seoul St. Mary's Hospital (Other); Kaohsiung Medical University (Other); Chang Gung Memorial Hospital (Other); E-DA Hospital (Other); Taitung Mackay Memorial Hospital (Unknown); National Cheng-Kung University Hospital (Other); Chi Mei Medical Hospital (Other); Chiayi Christian Hospital (Other); St. Martin De Porress Hospital (Other); Dalin Tzu Chi General Hospital (Other); Taichung Veterans General Hospital (Other); China Medical University Hospital (Other); Seoul National University Bundang Hospital (Other)
Responsible Party: Sponsor-Investigator, Young-Suk Lim, Professor, Asan Medical Center
Organization: Asan Medical Center (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IN-KR-320-5358
Record Dates: First submitted 2018-11-22; First posted 2018-11-26 (Actual); Last update posted 2024-12-17 (Actual); Status verified 2024-12

CONDITIONS: Chronic Hepatitis b
MeSH Terms: conditions — Hepatitis B, Chronic | interventions — tenofovir alafenamide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Treatment Arm A (TAF) (Experimental): 390 subjects administered Tenofovir Alafenamide 25 mg once daily
  Interventions: Drug: Tenofovir Alafenamide
- Treatment Arm B (Best supportive care) (No Intervention): 390 subjects received best supportive care
  During treatment period, among treatment arm B, subjects who are indicated for antiviral treatment will be treated with TAF as follows:
  1. Based on the AASLD 2018 Guidelines of CHB (ALT 70≥ for male, 50≥ for female)
  2. 40≤ALT levels<70 IU/L (males) or 40≤ ALT levels<50 IU/L (females) with evidence of significant fibrosis(F2; ≥7.2 kPa) as measured by either liver biopsy, Fibroscan or MR elastograpy performed within 3 months.
  3. If they were clinically judged to have cirrhosis by investigators and confirmed with Fibroscan (≥ 12.0 kPa).

INTERVENTIONS:
Drug: Tenofovir Alafenamide — Tenofovir Alafenamide 25mg, Tablet, Oral, Daily
  Other Names: Vemlidy
  Arms: Treatment Arm A (TAF)

SUMMARY:
Treatment with Tenofovir Alafenamide(TAF) in Chronic Hepatitis B (CHB) patients classified as beyond treatment indication of current international guidelines (e.g. aged more than 40 years old and 4 ≤ log HBV-DNA IU/mL < 8) is expected to bring improvement in long-term clinical outcomes. This expected result may expand the treatment indications in patients with CHB based on age and HBV-DNA in contrast to current international guidelines of CHB.

DETAILED DESCRIPTION:
Study objectives: To investigate whether TAF treatment reduce clinical events (HCC, death, liver decompensation, portal hypertensive complications, and liver transplantation) in CHB patients beyond treatment indications by current guidelines

Study procedure: 780 subjects will be randomized in a 1:1 ratio (A:B) either to receive TAF 25 mg QD or to receive best supportive care after stratification according to the HBeAg status.

The study duration is 12 years. During treatment period, among treatment arm B, subjects who are indicated for antiviral treatment will be treated with TAF as follows:

1. Based on the AASLD 2018 Guidelines of CHB (ALT 70≥ for male, 50≥ for female)
2. 40≤ALT levels<70 IU/L (males) or 40≤ ALT levels<50 IU/L (females) with evidence of significant fibrosis(F2; ≥7.2 kPa) as measured by either liver biopsy, Fibroscan or MR elastograpy performed within 3 months.
3. If they were clinically judged to have cirrhosis by investigators and confirmed with Fibroscan (≥ 12.0 kPa).

   * Treatment Arm A: 390 subjects administered TAF 25 mg once daily
   * Treatment Arm B: 390 subjects received best supportive care

The primary analysis will occur at Year 4 with the primary endpoint being occurrence of composite events during follow-up observation

ELIGIBILITY:
Inclusion Criteria: Patients must meet all of the following criteria to be eligible to participate in the study

1. Patient must have the ability to understand and sign a written informed consent form; consent must be obtained prior to initiation of study procedures
2. Male or female, 40 to 80 years of age
3. Positive for HBsAg or HBV DNA for at least 6 months or more
4. HBeAg positive or negative
5. No evidence of liver cirrhosis (platelet count ≥100,000/mm3)
6. serum HBV DNA ≥ 4 log10 IU/mL and ≤ 8 log10 IU/mL
7. Serum ALT level <70 if male, <50 if female
8. Estimated creatinine clearance ≥ 30 ml/min based on serum creatinine as measured at the screening evaluation
9. Patient is willing and able to comply with all study requirements

Exclusion Criteria: Patients who meet any of the following exclusion criteria are not to be enrolled in this study

1. Co-infection with HCV, HDV, HIV (Confirmed by nucleic acid tests)
2. Abusing alcohol (more than 60 g/day) or illicit drugs
3. Patients with history of hepatic decompensation (e.g., ascites, encephalopathy or variceal hemorrhage)

4-1) Evidence of cirrhosis, including any of follows:

1. Platelet count <100,000/mm3
2. Esophagogastric varices on endoscopy
3. Evidence of clinically significant portal hypertension
4. Fibroscan ≥ 12.0 kPa (If the test was done in 3 months before the time of screening.) and confirmed to have liver cirrhosis by an investigator

4-2) 40≤ALT levels<70 IU/L (males) or 40≤ ALT levels<50 IU/L (females) with evidence of significant fibrosis(F2; ≥7.2 kPa) as measured by either liver biopsy, Fibroscan or MR elastograpy performed within 3 months.

5. Received interferon or other immunomodulatory treatment for HBV infection in the 12 months before screening for this study

6. Medical condition that requires concurrent use of systemic corticosteroid or other immunosuppressive agents

7. Received solid organ or bone marrow transplant

8. Known hypersensitivity to study drugs, metabolites, or formulation excipients

9. Any other clinical condition or prior therapy that, in the opinion of the Investigator, would make the patient unsuitable for the study or unable to comply with dosing requirements

10. Use of investigational agents within 6 months of screening, unless allowed by the Sponsor or Investigator

11. Significant renal, cardiovascular, pulmonary, or neurological disease in the opinion of the Investigator

12. Any malignant tumor in the preceding five years. However, a history of treated malignancy (other than HCC) is allowable if the patient's malignancy has been in complete remission, off chemotherapy and without additional surgical intervention, during the preceding three years

13. Pregnant or breastfeeding or willing to be pregnant

14. Participating in other clinical trials to administer medication. However, it is possible to participate if it is not an antiviral agent or immunosuppressant related clinical trial.

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 780 (Estimated)
Dates: Start 2019-02-18 (Actual); Primary Completion 2031-12-31 (Estimated); Study Completion 2031-12-31 (Estimated)

PRIMARY OUTCOMES:
the occurrence of composite events during follow-up observation | At year 4
  the occurrence of composite events during follow-up observation(including death, liver transplantation, or decompensated liver diseases [Child-Pugh score≥7], complications of portal hypertension [ascites, gastroesophageal varices] or HCC

SECONDARY OUTCOMES:
Cumulative rate of patients with clinical events | At year 4, 8 and 12
  Cumulative rate of patients with clinical events (death, liver transplantation, liver decompensation, portal hypertensive complications, and HCC)
Cumulative incidence rate of HCC | At year 4, 8 and 12
  Cumulative incidence rate of HCC
All-cause mortality | At year 4, 8 and 12
  All-cause mortality
Cumulative incidence rate of liver transplantation | At year 4, 8 and 12
  Cumulative incidence rate of liver transplantation
Cumulative incidence rate of liver decompensation | At year 4, 8 and 12
  Cumulative incidence rate of liver decompensation
Cumulative incidence rate of portal hypertensive complications | At year 4, 8 and 12
  Cumulative incidence rate of portal hypertensive complications
Rate of receiving nucleos(t)ide analogue by meeting reimbursement criteria of treatment among Treatment ARM B subjects | At year 4, 8 and 12
  Rate of receiving nucleos(t)ide analogue by meeting reimbursement criteria of treatment among Treatment ARM B subjects
Virologic response defined as HBV DNA less than 15 IU/mL | At year 4, 8 and 12
  Virologic response defined as HBV DNA less than 15 IU/mL
Rate of ALT normalization | At year 4, 8 and 12
  Rate of ALT normalization if baseline ALT is elevated
Rate of HBeAg seroclearance and seroconversion | At year 4, 8 and 12
  Rate of HBeAg seroclearance and seroconversion among HBeAg-positive patients
Change of fibroscan | At year 4, 8 and 12
  Change of fibroscan
Change of APRI index | At year 4, 8 and 12
  Change of APRI index
Change of FIB-4 | At year 4, 8 and 12
  Change of FIB-4
Cumulative incidence rate of HCC among HBeAg-positive or HBeAg-negative Patients | At year 4, 8 and 12
  Cumulative incidence rate of HCC among HBeAg-positive or HBeAg-negative Patients
All cause-mortality among HBeAg-positive or HBeAg-negative | At year 4, 8 and 12
  All cause-mortality among HBeAg-positive or HBeAg-negative
Cumulative incidence rate of liver transplantation among HBeAg-positive or HBeAg-negative | At year 4, 8 and 12
  Cumulative incidence rate of liver transplantation among HBeAg-positive or HBeAg-negative
Cumulative incidence rate of liver decompensation among HBeAg-positive or HBeAg-negative | At year 4, 8 and 12
  Cumulative incidence rate of liver decompensation among HBeAg-positive or HBeAg-negative
Cumulative incidence rate of portal hypertensive complications among HBeAg-positive or HBeAg-negative | At year 4, 8 and 12
  Cumulative incidence rate of portal hypertensive complications amongHBeAg-positive or HBeAg-negative
Cumulative incidence rate of HCC among subjects according to baseline ALT level (normal ALT and elevated ALT) | At year 4, 8 and 12
  Cumulative incidence rate of HCC amongsubjects according to baseline ALT level (normal ALT and elevated ALT)
All cause-mortality among subjects according to baseline ALT level (normal ALT and elevated ALT) | At year 4, 8 and 12
  All cause-mortality among subjects according to baseline ALT level (normal ALT and elevated ALT)
Cumulative incidence rate of liver transplantation among subjects according to baseline ALT level (normal ALT and elevated ALT) | At year 4, 8 and 12
  Cumulative incidence rate of liver transplantation among subjects according to baseline ALT level (normal ALT and elevated ALT)
Cumulative incidence rate of liver decompensation among subjects according to baseline ALT level (normal ALT and elevated ALT) | At year 4, 8 and 12
  Cumulative incidence rate of liver decompensation among subjects according to baseline ALT level (normal ALT and elevated ALT)
Cumulative incidence rate of portal hypertensive complications among subjects according to baseline ALT level (normal ALT and elevated ALT) | At year 4, 8 and 12
  Cumulative incidence rate of portal hypertensive complications among subjects according to baseline ALT level (normal ALT and elevated ALT)
Cumulative and annual rate of patients with clinical events (death, liver transplantation, liver decompensation, portal hypertensive complications, and HCC) after excluding patients who occurrs clinical events within 6 months of enrollment | At year 4, 8 and 12
  Cumulative and annual rate of patients with clinical events (death, liver transplantation, liver decompensation, portal hypertensive complications, and HCC) after excluding patients who occurrs clinical events within 6 months of enrollment
Cumulative and annual rate of patients with clinical events (death, liver transplantation, liver decompensation, portal hypertensive complications, and HCC) after excluding patients who occurrs clinical events within 12 months of enrollment | At year 4, 8 and 12
  Cumulative and annual rate of patients with clinical events (death, liver transplantation, liver decompensation, portal hypertensive complications, and HCC) after excluding patients who occurrs clinical events within 12 months of enrollment
Cumulative and annual rate of patients with clinical events in patients with normal ALT (<40 U/L) at the time of enrollment, after excluding patients who occurrs clinical | At year 4, 8 and 12
  Cumulative and annual rate of patients with clinical events (death, liver transplantation, liver decompensation, portal hypertensive complications, and HCC) in patients with normal ALT (<40 U/L) at the time of enrollment, after excluding patients who occurrs clinical events within 6 months of enrollment
Cumulative and annual rate of patients with clinical events in patients with normal ALT (<40 U/L) at the time of enrollment, after excluding patients who occurrs clinical events within 12 months of enrollment | At year 4, 8 and 12
  Cumulative and annual rate of patients with clinical events (death, liver transplantation, liver decompensation, portal hypertensive complications, and HCC) in patients with normal ALT (<40 U/L) at the time of enrollment, after excluding patients who occurrs clinical events within 12 months of enrollment

CONTACTS AND LOCATIONS:
Overall Officials: Young-Suk Lim, M.D, Ph D, Principal Investigator — Asan Medical Center
Locations (10):
- South Korea (10):
  - Kyungpook National University Hospital, Daegu
  - Seoul National University Bundang Hospital, Seongnam
  - Asan Medical Center, Seoul
  - Chung-Ang University Hospital, Seoul
  - Konkuk University Hospital, Seoul
  - Korea University Guro Hospital, Seoul
  - Kyung-Hee University Hospital, Seoul
  - Samsung Medical center, Seoul
  - Seoul National University Hospital, Seoul
  - Ulsan University Hospital, Ulsan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Terrault NA, Lok ASF, McMahon BJ, Chang KM, Hwang JP, Jonas MM, Brown RS Jr, Bzowej NH, Wong JB. Update on prevention, diagnosis, and treatment of chronic hepatitis B: AASLD 2018 hepatitis B guidance. Hepatology. 2018 Apr;67(4):1560-1599. doi: 10.1002/hep.29800. No abstract available. PMID 29405329
- [Background] European Association for the Study of the Liver. EASL 2017 Clinical Practice Guidelines on the management of hepatitis B virus infection. J Hepatol. 2017 Aug;67(2):370-398. doi: 10.1016/j.jhep.2017.03.021. Epub 2017 Apr 18. PMID 28427875
- [Background] Tseng TC, Kao JH. Treating Immune-tolerant Hepatitis B. J Viral Hepat. 2015 Feb;22(2):77-84. doi: 10.1111/jvh.12370. Epub 2014 Nov 25. PMID 25424771
- [Background] Andreani T, Serfaty L, Mohand D, Dernaika S, Wendum D, Chazouilleres O, Poupon R. Chronic hepatitis B virus carriers in the immunotolerant phase of infection: histologic findings and outcome. Clin Gastroenterol Hepatol. 2007 May;5(5):636-41. doi: 10.1016/j.cgh.2007.01.005. Epub 2007 Apr 11. PMID 17428739
- [Background] Hui CK, Leung N, Yuen ST, Zhang HY, Leung KW, Lu L, Cheung SK, Wong WM, Lau GK; Hong Kong Liver Fibrosis Study Group. Natural history and disease progression in Chinese chronic hepatitis B patients in immune-tolerant phase. Hepatology. 2007 Aug;46(2):395-401. doi: 10.1002/hep.21724. PMID 17628874
- [Background] Kennedy PTF, Sandalova E, Jo J, Gill U, Ushiro-Lumb I, Tan AT, Naik S, Foster GR, Bertoletti A. Preserved T-cell function in children and young adults with immune-tolerant chronic hepatitis B. Gastroenterology. 2012 Sep;143(3):637-645. doi: 10.1053/j.gastro.2012.06.009. Epub 2012 Jun 15. PMID 22710188
- [Background] Lai M, Hyatt BJ, Nasser I, Curry M, Afdhal NH. The clinical significance of persistently normal ALT in chronic hepatitis B infection. J Hepatol. 2007 Dec;47(6):760-7. doi: 10.1016/j.jhep.2007.07.022. Epub 2007 Sep 24. PMID 17928090
- [Background] Kumar M, Sarin SK, Hissar S, Pande C, Sakhuja P, Sharma BC, Chauhan R, Bose S. Virologic and histologic features of chronic hepatitis B virus-infected asymptomatic patients with persistently normal ALT. Gastroenterology. 2008 May;134(5):1376-84. doi: 10.1053/j.gastro.2008.02.075. Epub 2008 Feb 29. PMID 18471514
- [Background] Kim GA, Lim YS, Han S, Choi J, Shim JH, Kim KM, Lee HC, Lee YS. High risk of hepatocellular carcinoma and death in patients with immune-tolerant-phase chronic hepatitis B. Gut. 2018 May;67(5):945-952. doi: 10.1136/gutjnl-2017-314904. Epub 2017 Oct 21. PMID 29055908
- [Background] Chen CJ, Yang HI, Su J, Jen CL, You SL, Lu SN, Huang GT, Iloeje UH; REVEAL-HBV Study Group. Risk of hepatocellular carcinoma across a biological gradient of serum hepatitis B virus DNA level. JAMA. 2006 Jan 4;295(1):65-73. doi: 10.1001/jama.295.1.65. PMID 16391218
- [Background] Iloeje UH, Yang HI, Su J, Jen CL, You SL, Chen CJ; Risk Evaluation of Viral Load Elevation and Associated Liver Disease/Cancer-In HBV (the REVEAL-HBV) Study Group. Predicting cirrhosis risk based on the level of circulating hepatitis B viral load. Gastroenterology. 2006 Mar;130(3):678-86. doi: 10.1053/j.gastro.2005.11.016. PMID 16530509
- [Background] Lin ZH, Xin YN, Dong QJ, Wang Q, Jiang XJ, Zhan SH, Sun Y, Xuan SY. Performance of the aspartate aminotransferase-to-platelet ratio index for the staging of hepatitis C-related fibrosis: an updated meta-analysis. Hepatology. 2011 Mar;53(3):726-36. doi: 10.1002/hep.24105. Epub 2011 Feb 11. PMID 21319189
- [Background] Sterling RK, Lissen E, Clumeck N, Sola R, Correa MC, Montaner J, S Sulkowski M, Torriani FJ, Dieterich DT, Thomas DL, Messinger D, Nelson M; APRICOT Clinical Investigators. Development of a simple noninvasive index to predict significant fibrosis in patients with HIV/HCV coinfection. Hepatology. 2006 Jun;43(6):1317-25. doi: 10.1002/hep.21178. PMID 16729309
- [Derived] Lim YS, Yu ML, Choi J, Chen CY, Choi WM, Kang W, Kim GA, Kim HJ, Lee YB, Lee JH, Park NH, Kwon SY, Park SY, Kim JH, Choi GH, Jang ES, Chen CH, Hsu YC, Bair MJ, Cheng PN, Tung HD, Chang TS, Lo CC, Tseng KC, Yang SS, Peng CY, Han S. Early antiviral treatment with tenofovir alafenamide to prevent serious clinical adverse events in adults with chronic hepatitis B and moderate or high viraemia (ATTENTION): interim results from a randomised controlled trial. Lancet Gastroenterol Hepatol. 2025 Apr;10(4):295-305. doi: 10.1016/S2468-1253(24)00431-X. Epub 2025 Feb 3. PMID 39914435

DOCUMENTS (2):
  • Study Protocol (2023-09-26): https://cdn.clinicaltrials.gov/large-docs/74/NCT03753074/Prot_000.pdf
  • Statistical Analysis Plan (2023-09-26): https://cdn.clinicaltrials.gov/large-docs/74/NCT03753074/SAP_001.pdf